CLINICAL TRIAL: NCT03484156
Title: Predictive Platform for PEople aGed and Requiring ASsistancE
Acronym: 3PEGASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/15/7803
Record Dates: First submitted 2017-06-15; First posted 2018-03-30 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Aging
Keywords: Elderly; Frailty; Tele-monitoring; Disability
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers (Experimental): The Installation of 3PEGASE Sensor in elders volunteers to monitor clinical indicators at home.The instrument is for monitoring functional and cognitive autonomy in frail or disable elderly persons living alone at home.
  The volunteers will have 70 years old or more, living alone at home, frail of disable (ADL> or =3) and able to walk by themselves.
  Interventions: Device: Installation of 3PEGASE Sensor

INTERVENTIONS:
Device: Installation of 3PEGASE Sensor — Volunteers will be equipped with the 3-PEGASE solution to monitor clinical indicators at home : By assessing older person's autonomy at home and detecting early infra-clinical indicators, the solution could provide relevant clinical parameters to the caregivers and healthcare professionals in order to support the patient's follow-up, and support the detection of preliminary signs of functional loss

SUMMARY:
The study aim is to assess the capacity of a technological solution for analyzing older person's functional and cognitive autonomy at home. Results from this study will also be used to elaborate the design of a further larger national multicenter randomized control trial assessing the efficacy of the solution to detect early infra-clinical disability.

DETAILED DESCRIPTION:
The object of the present project is to evaluate an instrument for monitoring functional and cognitive autonomy in frail or disable elderly persons living alone at home. By assessing older person's autonomy at home and detecting early infra-clinical indicators, the solution could provide relevant clinical parameters to the caregivers and healthcare professionals in order to support the patient's follow-up, and support the detection of preliminary signs of functional loss. The device consists of a set of sensors embedded in the house with minimal invasiveness. The solution transmits the collected data to a remote storage server. Data will then be available for distance consultations by users (i.e., patients, careers or physicians). The study will conduct a wide range of evaluations of the device (technical, clinical, and economic), which will allow the optimization of the prototype. The evaluation of the solution will involve 25 frail or disable community-dwelling subjects living alone for 6 months. Comprehensive assessments will be conducted to highlight the feasibility, integration in healthcare network, and clinical relevance of the technological device.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 75 or more, living alone at home
* frail of disable (ADL superior or equal at 3)
* able to walk by themselves

Exclusion Criteria:

* patient presenting a Mini Mental State lower at 16/30 and without a daily intervention from a caregiver
* non agreement of study participation of patients or the reliable person when appropriate.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
The occurrence of alerts | 6 months
  The occurrence of alerts : each alert will be recorded to characterize the number and the pace of alerts during the time of follow-up

SECONDARY OUTCOMES:
The relevance of each alert according to the subjective opinion | 6 months
  The relevance of each alert if it's legitimate or not legitimate according to the subjective opinion of ; the investigator and the voluntary subject The "Classic" alerts (volunteers on behalf of the person being followed) generated by the system will be defined as valid or invalid on the basis of the carers' assessment: "was he legitimate to alert you? And professionals (assistance).
  The "automatic" alerts generated by the sensors will be defined as valid or not on the basis of the assessment of the tele-assistant, the carer and the voluntary subject.

OTHER OUTCOMES:
The occurrence of major clinical events | 6 months
  The occurrence of major clinical events collected by the Clinical Research Assistant every 2 months a clinical event that required to bring in a doctor, firefighters, a call to 15 or at SOS doctor, a transport to an emergency service
The functional autonomy | 6 months
  The functional autonomy measured every 2 months by the Activities of Daily Living (ADL) score
The cognitive autonomy | 6 months
  The cognitive autonomy measured every two months by the Mini Mental State Examination (MMSE) score

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Piau, MD, Principal Investigator — Toulouse CHU
Locations (2):
- France (2):
  - University Hospital, Toulouse, Toulouse, Midi-Pyrenes
  - CHU Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piau A, Lepage B, Bernon C, Gleizes MP, Nourhashemi F. Real-Time Detection of Behavioral Anomalies of Older People Using Artificial Intelligence (The 3-PEGASE Study): Protocol for a Real-Life Prospective Trial. JMIR Res Protoc. 2019 Nov 18;8(11):e14245. doi: 10.2196/14245. PMID 31738180